CLINICAL TRIAL: NCT07357792
Title: Effectiveness of a Randomized Complex Intervention With Adolescents and Their Environment to Assess the Reduction of Problematic Video Game Use and Potential Video Game Addiction by Promoting Shared Active Leisure and Personal Development
Brief Title: Community-based Study With 1st-year Secondary Students (n=1104) and Their Environment. It Evaluates a Complex Intervention (Community Actions, Classroom-based Mindfulness for Adolescents, and Online Mindfulness for Adults) to Reduce Problematic Video Game Use and Improve Well-being.
Acronym: AQJ
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AQUÉJUGAMOS 2025/317
Record Dates: First submitted 2025-12-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Video Game Addiction; Gaming Disorder
Keywords: gaming disorder; video game addiction; mindfulness; social support; cyberbullying; impulsivity; well-being
MeSH Terms: conditions — Technology Addiction; Cyberbullying; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: This is a community-based, non-blinded, controlled interventional study with parallel groups. Allocation is performed at the classroom level within participating schools. The study uses a longitudinal design with repeated measurements (pre-intervention, post-intervention, and follow-up) to assess the effectiveness of a multi-component intervention implemented under real-world conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this arm include adolescents enrolled in the first year of secondary education from schools assigned to the intervention group, as well as adults from their close environment. Adolescents receive a complex, multi-component intervention consisting of a community-based component promoting active, shared, and screen-free leisure, and a classroom-based mindfulness and emotional development program. Adults from the adolescents' environment (family members and selected community, educational, and health professionals) participate in an individual, online mindfulness and emotional regulation program. All components are implemented in addition to usual school activities.
  Interventions: Behavioral: Community-Based Participatory Leisure Intervention; Behavioral: Classroom-Based Mindfulness and Emotional Development Program (Adolescents); Behavioral: Online Mindfulness and Emotional Regulation Program (Adults)
- Control Group (No Intervention): Participants in this arm include adolescents enrolled in the first year of secondary education from schools assigned to the control group. These participants do not receive any of the intervention components and continue with usual school activities. They participate only in data collection at the predefined assessment time points.

INTERVENTIONS:
Behavioral: Community-Based Participatory Leisure Intervention — This intervention consists of a community-based component designed to promote active, shared, and screen-free leisure among adolescents. It is implemented through the creation of a school-based community group composed of adolescents, teachers, health professionals, family representatives, and community members. Adolescents actively participate in identifying community leisure resources, co-designing leisure activities, and implementing and disseminating these activities within their local environment using participatory action research methodologies.
  Arms: Intervention Group
Behavioral: Classroom-Based Mindfulness and Emotional Development Program (Adolescents) — This intervention is a structured, classroom-based mindfulness and emotional development program delivered to adolescents during school hours. The program is based on established mindfulness protocols and consists of multiple sessions aimed at improving attention, emotional awareness, stress management, and self-regulation. Sessions combine experiential mindfulness practices, reflective activities, and group discussions adapted to early adolescence.
  Arms: Intervention Group
Behavioral: Online Mindfulness and Emotional Regulation Program (Adults) — This intervention is an individual, self-guided online program for adults from the adolescents' environment, including family members and selected educational, health, and community professionals. The program combines mindfulness practices and cognitive-behavioral strategies to improve emotional regulation, stress management, and well-being, and to strengthen adults' capacity to support adolescents in developing healthy leisure habits.
  Arms: Intervention Group

SUMMARY:
The goal of this observational, community-based study is to evaluate the effectiveness of a complex intervention designed to reduce problematic video game use and the risk of video game addiction in adolescents, while promoting active, shared leisure activities and personal and emotional development.

The study involves students in the first year of secondary education (approximately 12-13 years old) from multiple schools in Pontevedra (Galicia, Spain), as well as adults from their close environment, including family members, teachers, health professionals, and community representatives. Schools are assigned either to an intervention group or to a control group with similar sociodemographic characteristics.

The study is based on a systems and community perspective, assuming that adolescents' video game use is influenced by individual factors (such as impulsivity and emotional regulation), as well as by family, school, and community contexts and the availability of appealing leisure alternatives. For this reason, the intervention consists of three coordinated components that are implemented over time in the intervention schools.

The main questions the study aims to answer are: (a) Can a complex intervention combining community participation and mindfulness-based training reduce problematic video game use and the risk of video game addiction in adolescents?; (b) Does classroom-based mindfulness training improve adolescents' mindfulness, emotional well-being, and self-regulation?; (c) Does mindfulness training for adults improve their own well-being and their ability to support adolescents in adopting healthier leisure habits?; and (d) Can a participatory, community-based approach increase adolescents' awareness and use of active, screen-free leisure alternatives?

Researchers will compare adolescents from intervention schools with adolescents from control schools, where no intervention is implemented and only data are collected. Outcomes will be measured at three time points: before the intervention, after the intervention, and at follow-up, in order to assess changes over time and the sustainability of effects.

Participants will:

* Complete questionnaires at different time points assessing video game use, possible video game addiction, mindfulness, psychological well-being, impulsivity, cyberbullying, social support, and online experiences.
* Take part in a community-based component in which adolescents actively participate in identifying, designing, and promoting leisure activities without screens in their local environment. This process includes the creation of a school-based community group composed of adolescents, teachers, health professionals, family representatives, and community members. Adolescents are involved in participatory activities to map community resources and co-design attractive leisure options, which are later implemented and shared with families and the wider community.
* Participate in a group-based mindfulness and emotional development program delivered in the classroom during school hours. This program consists of structured sessions based on established mindfulness protocols and is designed to help adolescents develop attention skills, emotional awareness, stress management, and self-regulation.
* Access an individual, online mindfulness and emotional regulation program (adults only), which combines mindfulness practices and cognitive-behavioral strategies. This self-guided program is completed over several weeks and aims to improve adults' well-being and provide tools to better support adolescents.

By integrating community action, school-based intervention, and adult involvement, this study seeks to evaluate a comprehensive and sustainable approach to preventing problematic video game use and promoting healthier lifestyles during adolescence

DETAILED DESCRIPTION:
Video games are a common form of leisure among adolescents and can have positive effects when used in moderation. However, excessive or problematic use during adolescence has been associated with negative consequences for physical health, emotional well-being, academic performance, and social relationships. In recent years, concerns have increased regarding the risk of problematic video game use and potential video game addiction, particularly in relation to online gaming, prolonged screen time, and difficulties in emotional self-regulation.

Adolescence is a critical developmental period in which habits related to leisure, coping strategies, and emotional regulation are established. Research suggests that problematic video game use does not depend solely on individual behavior, but is influenced by a combination of personal, family, school, and community factors.

The widespread use of video games among adolescents has increased substantially in recent years, making digital gaming one of the main forms of leisure during this developmental stage. While video games can offer entertainment and social interaction, research has shown that excessive or poorly regulated use may be associated with sedentary behavior, sleep disturbances, emotional difficulties, academic problems, and impaired social relationships. In response to these concerns, problematic video game use has been increasingly examined as a public health and mental health issue in adolescence.

The present study is grounded in current scientific evidence indicating that problematic video game use is influenced by multiple interacting factors. These include individual characteristics such as impulsivity, emotional regulation, and stress, as well as contextual factors related to family functioning, school environment, community resources, and the design features of contemporary video games. The study also draws on evidence supporting mindfulness-based approaches as promising tools for improving self-control, emotional awareness, and well-being in adolescents and adults.

The study follows a longitudinal, controlled design with an intervention group and a control group. Participating schools are located in different basic health zones in Pontevedra (Galicia, Spain), representing urban, semi-urban, rural, and coastal contexts. Schools in the intervention and control groups are selected to ensure comparable sociodemographic characteristics.

Allocation is performed at the classroom level, and blinding of participants is not feasible due to the nature of the intervention. However, blinding is applied during data analysis. The study is embedded within the official school planning framework, facilitating institutional support and high participation rates.

The planned sample includes approximately 1,104 adolescents, with 552 students in the intervention group and 552 in the control group. Sample size calculations are based on detecting a 35% reduction in problematic video game use and potential video game addiction, assuming an initial prevalence of approximately 18%. Calculations were performed using standard epidemiological software.

In addition to adolescents, the study includes adults from the adolescents' environment, such as family members, teachers, health professionals, and community representatives, who participate in specific components of the intervention.

The intervention is structured around three coordinated components: a community-based component, a group-based component for adolescents, and an individual component for adults. These components are implemented sequentially and are designed to reinforce each other.

The community-based component aims to promote active, shared, and screen-free leisure activities within the adolescents' local environment. A central element is the creation of a school-based community group composed of adolescents, teachers, health professionals, family representatives, and community members.

This group is trained in participatory action research methodologies, enabling adolescents to actively identify community assets, barriers, and opportunities related to leisure activities. Adolescents participate in mapping local resources, prioritizing feasible and attractive alternatives to video gaming, and co-designing leisure activities adapted to their context.

The selected activities are implemented through organized community events and leisure sessions, which may include physical, recreational, or volunteer activities. Dissemination activities are conducted to share experiences and outcomes with families, schools, health services, and the broader community. This component emphasizes adolescent leadership, shared decision-making, and sustainability.

The group-based component consists of a classroom-based mindfulness and emotional development program delivered to adolescents in intervention schools. The program is based on internationally recognized mindfulness protocols and is adapted to the educational context and developmental stage of early adolescence.

The program is delivered through structured sessions during school hours, focusing on the development of attention, emotional awareness, stress management, and self-regulation. Sessions combine experiential practices, reflective activities, and age-appropriate discussions. No minimum number of participants is required, and adaptations are made to ensure accessibility for students with special educational needs.

This component is designed to address individual factors associated with problematic video game use, such as impulsivity and emotional dysregulation, while complementing the community-based activities.

The individual component targets adults from the adolescents' environment, including family members and members of the community group. It consists of an online, self-guided program combining mindfulness practices and cognitive-behavioral strategies.

The program is delivered through digital platforms and completed over several weeks. It includes structured modules with guided practices, psychoeducational content, and exercises aimed at improving emotional regulation, stress management, and well-being. Participation is voluntary and requires informed consent.

This component is intended to strengthen the supportive role of adults and to promote consistency between adolescents' environments, reinforcing healthy leisure habits and emotional skills.

Data are collected at three time points: baseline (pre-intervention), post-intervention, and follow-up. Validated instruments are used to assess problematic video game use, potential video game addiction, mindfulness, psychological well-being, impulsivity, cyberbullying, social support, and online experiences. Adult participants complete measures related to mindfulness.

Adherence to each intervention component is systematically recorded using attendance logs and digital access records, allowing assessment of engagement and dose-response relationships.

Data are managed using a secure electronic data capture system with pseudonymization and separation of identifying information. This ensures compliance with data protection regulations and supports data integrity.

Statistical analyses are conducted using multilevel mixed-effects models to account for the hierarchical structure of the data (students nested within classrooms and schools) and repeated measurements over time. Analyses compare changes between intervention and control groups while adjusting for relevant covariates such as age, sex, adherence, and contextual factors.

Predefined criteria for intervention success are established based on relative improvements in primary and secondary outcomes, informed by the absence of closely comparable prior interventions.

The study complies with ethical principles for research involving minors, including informed consent procedures and special protections for confidentiality and inclusion. Activities are adapted to ensure accessibility for participants with special educational needs.

Dissemination is integrated throughout the study, with structured activities aimed at families, schools, health services, and the community. Study data are prepared following FAIR principles to support transparency and future research.

ELIGIBILITY:
Inclusion Criteria:

* FOR ADOLESCENTS:
* Age between 11 and 15 years at the time of enrollment.
* Enrollment in the first year of secondary education in a participating school.
* Attendance in a classroom assigned to either the intervention or control group.
* Provision of written informed consent by a parent or legal guardian.
* Provision of assent by the adolescent, when applicable according to age and regulations (14 years old).
* FOR ADULTS:
* Being a parent, legal guardian, teacher, health professional, or community member linked to an adolescent in the intervention group.
* Willingness to participate in the adult component of the study.
* Provision of written informed consent.

Exclusion Criteria:

* FOR ADOLESCENTS:
* Age below 11 years or above 15 years at the time of enrollment.
* Lack of written informed consent from a parent or legal guardian.
* Refusal or inability of the adolescent to provide assent, when applicable.
* Inability to complete the study questionnaires due to language or comprehension barriers that cannot be reasonably accommodated.
* FOR ADULTS:
* Lack of written informed consent.
* Inability to access or use the digital platform required for the online intervention.
* Inability to complete study questionnaires due to language or comprehension barriers.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1668 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Problematic Video Game Use and Potential Video Game Addiction | One year and at follow-up (6 months after study completion)
  Change in problematic video game use and potential video game addiction among adolescents, assessed using validated self-report instruments. Outcomes are measured through the Game Addiction Scale for Adolescents and the Ten-Item Internet Gaming Disorder Test. The minimum score of the Game Addiction Scale for Adolescents is 7 and the maximum score is 35; higher scores indicate greater severity of problematic use or addiction-related symptoms. The minimum score of the Ten-Item Internet Gaming Disorder Test is 0 and the maximum score is 10; higher scores indicate greater serverity of problematic use or addiction-related symptoms.

SECONDARY OUTCOMES:
Mindfulness in Adolescents | One year and at follow-up (6 months after study completion)
  Change in mindfulness levels among adolescents, assessed using the Child and Adolescent Mindfulness Measure. The scale evaluates attention to the present moment and acceptance of internal experiences. The minimum score is 5 and the maximum 25; higher scores indicate higher and better levels of mindfulness.
Psychological Well-Being in Adolescents | One year and at follow-up (6 months after study completion)
  Change in psychological well-being among adolescents, assessed using the Psychological Well-Being Scale for Children and Adolescents, which measures multiple dimensions of well-being. The minimum score is 6 and the maximum is 36; higher scores indicate higher and better levels of mindfulness.
Impulsivity in Adolescents | One year and at follow-up (6 months after study completion)
  Change in impulsivity traits among adolescents, assessed using the Scale of Impulsivity for Children and Adolescents. This scale consists of five subscales that are scored individually using Likert-type responses ranging from 1 to 4. The minimum score for the "Negative Urgency," "Sensation Seeking," and "Positive Urgency" subscales is 4 and the maximum is 16; higher scores indicate greater impulsivity. The remaining two subscales have the same minimum and maximum scores but are composed entirely of reverse-scored items; higher scores indicate greater lack of perseverance and lack of premeditation.
Cyberbullying Involvement | One year and at follow-up (6 months after study completion)
  Prevalence and change in involvement in cyberbullying behaviors among adolescents, assessed using the Spanish version of the European Cyberbullying Intervention Project Questionnaire, which consists of 22 Likert-type items with response options scored from 0 to 4. It comprises two dimensions: cybervictimization and cyberaggression. The minimum score for each dimension is 11 and the maximum is 44; higher scores indicate greater involvement in the cyberbullying phenomenon, either as a victim or as a perpetrator.
Perceived Social Support | One year and at follow-up (6 months after study completion)
  Change in perceived social support among adolescents, assessed using the Multidimensional Scale of Perceived Social Support, which consists of 12 items measuring perceived adequacy of social support from three sources: family members, friends, and significant others. These 12 items are rated on a 7-point Likert-type scale ranging from 1 to strongly agree 7. The minimum score is 12 and the maximum score is 84. The total score corresponds to the sum of the scores for each item, with higher or lower scores indicating greater or lesser perceived social support, respectively.
Self-Reported Video Game Use Time | One year and at follow-up (6 months after study completion)
  Change in the number of hours spent playing video games, self-reported by adolescents using an ad hoc questionnaire.
Mindfulness in Adults | One year and at follow-up (6 months after study completion)
  Change in mindfulness levels among adults from the adolescents' environment, assessed using the Five Facets of Mindfulness Questionnaire. Consists of 15 Likert-type items with five response options ([1] "Never or very rarely true" to [5] "Always or almost always true") and assesses five dimensions of mindfulness: observing, describing, acting with awareness, nonjudging of inner experience, and nonreactivity to inner experience. The minimum score is 15 and the maximum score is 75; higher scores indicate higher and greater levels of mindfulness.
Family-Reported Video Game Use | At the start of the intervention, with a maximum duration of 6 months.
  Change in the number of hours spent playing video games as reported by family members of adolescents in the intervention group, collected using an ad hoc questionnaire.

OTHER OUTCOMES:
Adherence to the Community Component | Throughout the intervention period (an average of 1 year).
  Level of adherence to the community-based intervention component, assessed through systematic attendance records of participation in community sessions and activities.
Adherence to the Group-Based Mindfulness Program (Adolescents) | Throughout the intervention period (an average of 1 year).
  Level of adherence to the classroom-based mindfulness and emotional development program, measured by attendance records across scheduled sessions.
Adherence to the Individual Online Program (Adults) | Throughout the intervention period (an average of 8 months).
  Level of adherence to the individual online mindfulness and emotional regulation program for adults, assessed through automated platform access and activity logs.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Clavería Fontán, Primary Care Health Technician, Principal Investigator — Servicio Gallego de Salud
Locations (1):
- Centro de Saúde de Rosalía de Castro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mettler, J., Mills, D.J., Heath, N.L. (2020). Problematic Gaming and Subjective Well-Being: How Does Mindfulness Play a Role? International Journal of Mental Health and Addiction, 18(3), 720-736.
- [Background] Kim J, Lee S, Lee D, Shim S, Balva D, Choi KH, Chey J, Shin SH, Ahn WY. Psychological treatments for excessive gaming: a systematic review and meta-analysis. Sci Rep. 2022 Nov 28;12(1):20485. doi: 10.1038/s41598-022-24523-9. PMID 36443408
- [Background] Ji Y, Yin MXC, Zhang AY, Wong DFK. Risk and protective factors of Internet gaming disorder among Chinese people: A meta-analysis. Aust N Z J Psychiatry. 2022 Apr;56(4):332-346. doi: 10.1177/00048674211025703. Epub 2021 Jul 10. PMID 34250835
- [Background] Király, O., Griffiths, M.D., & Demetrovics, Z. (2015). Internet Gaming Disorder and the DSM-5: Conceptualization, Debates, and Controversies. Current Addiction Reports, 2(3), 254-262.
- [Background] King DL, Delfabbro PH, Billieux J, Potenza MN. Problematic online gaming and the COVID-19 pandemic. J Behav Addict. 2020 Apr 29;9(2):184-186. doi: 10.1556/2006.2020.00016. Print 2020 Jun. PMID 32352927
- [Background] Andrade-Pérez, B.A., Guadix-García, I.G., Rial-Boubeta, A.R., & Suárez-Lorenzo, F.S. (2021). El impacto de la tecnología en la adolescencia: relaciones, riesgos y oportunidades. UNICEF.
- [Background] Gao YX, Wang JY, Dong GH. The prevalence and possible risk factors of internet gaming disorder among adolescents and young adults: Systematic reviews and meta-analyses. J Psychiatr Res. 2022 Oct;154:35-43. doi: 10.1016/j.jpsychires.2022.06.049. Epub 2022 Jul 19. PMID 35926424
- [Background] Derevensky JL, Hayman V, Lynette Gilbeau. Behavioral Addictions: Excessive Gambling, Gaming, Internet, and Smartphone Use Among Children and Adolescents. Pediatr Clin North Am. 2019 Dec;66(6):1163-1182. doi: 10.1016/j.pcl.2019.08.008. PMID 31679605
- [Background] Rial Boubeta, A. R. (2022). Adolescencia, tecnología, salud y convivencia: un estudio integral y proactivo desde los propios adolescentes. Fundación Barrié.